CLINICAL TRIAL: NCT03392467
Title: A Multi-center, Randomized, Double-blind, Parallel, Placebo-controlled Phase II Clinical Trial to Evaluate the Efficacy and Safety of PNEUMOSTEM for the Prevention and Treatment of Severe Bronchopulmonary Dysplasia in Premature Infants
Brief Title: PNEUMOSTEM for the Prevention and Treatment of Severe BPD in Premature Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medipost Co Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MP-CR-012
Record Dates: First submitted 2017-12-20; First posted 2018-01-08 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-03

CONDITIONS: Severe Bronchopulmonary Dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNEUMOSTEM (Experimental): human umbilical cord blood derived mesenchymal stem cell (hUCB-MSC)
  Interventions: Biological: PNEUMOSTEM
- Placebo (Placebo Comparator): normal saline
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: PNEUMOSTEM — human umbilical cord blood-derived mesenchymal stem cells
  Arms: PNEUMOSTEM
Other: Placebo — normal saline
  Arms: Placebo

SUMMARY:
This study is to evaluate the efficacy and safety of PNEUMOSTEM® for the Prevention and Treatment of Severe Bronchopulmonary Dysplasia (Severe BPD) in Premature Infants. Half of subjects will receive PNEUMOSTEM, while the other half will receive a placebo.

DETAILED DESCRIPTION:
Bronchopulmonary dysplasia (BPD) is a chronic lung disease in which premature infants and it results in significant morbidity and mortality. PNEUMOSTEM is intended to prevent and treat BPD by modulating inflammation and repairing damaged lung tissue in premature infants through paracrine effects.

ELIGIBILITY:
Inclusion Criteria:

at screening and randomization

1. 23 weeks to < 25 weeks of gestational age
2. 500g to 1,250g body weight at birth
3. premature infant within postnatal 13 days of age
4. use ventilator with ventilation rate >12 breaths/min or oxygen supply > 25%, or use high frequency ventilator (HFV)

at IP administration

1. premature infant within postnatal 5 to 14 days of age
2. No improvement in ventilator setting 24 hours prior to administration of IP

Exclusion Criteria:

1. subject with cyanotic congenital heart disease or non-cyanotic congenital heart disease that can cause heart failure
2. subject with pulmonary hypoplasia, congenital diaphragmatic hernia, or serious lung malformation such as congenital cystic lung disease
3. subject with chromosome disorder with serious malformation (i.e. Edward syndrome, patau syndrome, Down syndrome, etc.), severe congenital malformation (i.e. hydrocephalus, encephalocele, etc.), or severe congenital infection (i.e., herpes, toxoplasmosis, rubella, syphilis, AIDS, etc.)
4. subject with serious sepsis as active infection or shock due to sepsis
5. subject with grade 3 or 4 of bilateral intraventricular hemorrhage
6. at screening, subject with active pulmonary hemorrhage or active air leak syndrome
7. subject who underwent/will undergo surgery within 72 hours before/after investigational product (IP) administration
8. subject who is expected to be treated with surfactant within 24 hours prior to IP administration
9. subject who is expected to be allergic to gentamicin (Birth mother's allergy for gentamicin will be confirmed).
10. subject who have previously participated in other clinical trials
11. subject who is considered ineligible by investigator due to other medical reasons

Max Age: 13 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects who have severe BPD or are dead | 36 weeks postmenstrual age (PMA)
  Percentage of subjects who have severe BPD or are dead

SECONDARY OUTCOMES:
Percentage of subjects who have moderate/severe BPD or are dead | 36 weeks PMA
  Percentage of subjects who have moderate/severe BPD or are dead
Percentage of subjects by severity of BPD | prenatal 28 days/36 weeks PMA
  Percentage of subjects by severity of BPD
Percentage of subjects in death due to lung disease | prenatal 28 days/36 weeks PMA and study end timepoint
  Percentage of subjects in death due to lung disease
intubation duration | up to 24 weeks
  intubation duration
ventilation duration | up to 24 weeks
  ventilation duration
continuous positive airway pressure (CPAP) treatment duration | up to 24 weeks
  continuous positive airway pressure (CPAP) treatment duration
treatment duration with supplemental oxygen | up to 24 weeks
  treatment duration with supplemental oxygen
% of subjects treated with steroid for weaning ventilator | up to 24 weeks
  % of subjects treated with steroid for weaning ventilator
Retinopathy of prematurity (ROP) with stage III or higher | up to 24 weeks
  number of subjects with ROP with stage III or higher
number of subjects with retinopathy of prematurity that needs bevacizumab or laser therapy | up to 24 weeks
  number of subjects with retinopathy of prematurity that needs bevacizumab or laser therapy
z-score | up to 24 weeks (visit 10)
  percentile for body weight, height, and head circumference
days in hospitalization | up to 24 weeks
  days in hospitalization
changes in tracheal suction fluid examination | from screening to 7 days after IP administration (visit 5)
  changes in tracheal suction fluid examination

CONTACTS AND LOCATIONS:
Overall Officials: Wonsoon Park, Principal Investigator — Samsung Medical Center; Airhan Kim, Principal Investigator — Asan Medical Center
Locations (2):
- South Korea (2):
  - Asan medical Center, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ahn SY, Chang YS, Lee MH, Sung SI, Lee BS, Kim KS, Kim AR, Park WS. Stem cells for bronchopulmonary dysplasia in preterm infants: A randomized controlled phase II trial. Stem Cells Transl Med. 2021 Aug;10(8):1129-1137. doi: 10.1002/sctm.20-0330. Epub 2021 Apr 20. PMID 33876883